CLINICAL TRIAL: NCT06558734
Title: Evaluation of the Clinical Success of Pediatric Fiberglass Crowns in Primary Teeth Using Different Luting Cements
Brief Title: Pediatric Fiberglass Crown in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Zulfikar Zahit Ciftci, Head of Principal Dentisty, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDH-2020-5280
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries; Dental Plaque
Keywords: Fiberglass crown; Glass-ionomer cement; Resin-modified glass-ionomer cement; Primary molar teeth
MeSH Terms: conditions — Dental Caries; Dental Plaque | interventions — Cementation

STUDY DESIGN:
Who Masked: Participant
Masking Description: The treatments and evaluations were conducted by different researchers. As a result, masking could be performed for both the investigators and the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device: Glass-ionomer cement (Experimental): The capsule was attached to the mixer and mixed for 10 seconds. The cement was evenly distributed to the crowns paying attention that there were no air voids. Then crowns were placed by pressing them onto the prepared teeth with finger pressure. At least 2 minutes and 15 seconds after mixing, the excess cement was cleaned off. Following mixing, a minimum of 4 minutes and 30 seconds was allowed for the cement to set.
  Interventions: Procedure: Tooth Preperation; Procedure: Cementation
- Device: Resin-modified glass-ionomer cement (Experimental): FujiCEM 2 (GC, Tokyo, Japan) was evenly distributed to the inner surface of the crown with the syringe and immediately placed onto the teeth with finger pressure. The crowns were placed on the prepared tooth. At least 2 minutes and 15 seconds after mixing, the excess cement was cleaned off. Following mixing, a minimum of 4 minutes and 30 seconds was allowed for the cement to set.
  Interventions: Procedure: Tooth Preperation; Procedure: Cementation

INTERVENTIONS:
Procedure: Tooth Preperation — After the caries were removed, the teeth were prepared according to the manufacturer's recommendations for Figaro Crowns. Fiberglass crowns (Figaro Crowns Inc., USA) of the most suitable size in terms of the mesio-distal dimension of the tooth were selected. Following the establishment of anesthesia, the teeth were prepared using diamond cutting burs with a high-speed, water-cooled turbine handpiece. In order to achieve adequate interocclusal space, an occlusal reduction of 1-2 mm was executed along with a proximal reduction reaching 1 mm below the gingival margin. A more conservative reduction was applied to the buccal and lingual surfaces. After preparation, any remaining decayed dentin tissue was removed using a steel round bur with a low-speed micromotor. To ensure occlusal harmony, diamond burs were used to perform abrasion on the crown edges, and the trimmed crown edges were polished using rubber aids before cementation.
Procedure: Cementation — Figaro crowns were placed on the prepared teeth with finger pressure, following the manufacturer's instructions for the luting cement to be used. For each cement, the recommended setting time was observed, and excess cement residues were removed accordingly.

SUMMARY:
This randomized controlled clinical trial aims to evaluate the clinical success of fiberglass crowns applied to primary teeth and to assess the impact of two different luting cements on the success of the fiberglass crowns. The main questions to answer are:

* Will fiberglass crowns demonstrate sufficient clinical success to serve as a viable alternative to existing pediatric crowns?
* Will there be any differences in the clinical success and mechanical properties of fiberglass crowns based on the type of luting cement used?

Thirty-eight children (60 teeth), between 5 and 9 years old (7.03±1.14), enrolled for the study. The researchers evaluated the clinical success of fiberglass crowns bonded with two different types of luting cement (1: FujiOne; 2: FujiCEM 2) based on retention, anatomical integrity, effect on periodontal health and parental satisfaction.

Participants will:

-Visit the clinic 1st, 3rd, 6th, 12th months after cementatiton.

ELIGIBILITY:
Inclusion Criteria:

For participants:

* absence of any systemic disease
* absence of any periodontal disease
* no unilateral chewing habit
* a Frankl scale score of three-four

For teeth:

* no percussion or palpation sensitivity
* no malocclusion
* no pathological mobility
* no pulpal treatment due to caries or other reasons
* had sound cervical margins
* not hypoplastic or hypocalcified
* had opposing functioning teeth
* had physiological root resorption not exceeding one-third of the root length
* had deep dentin caries with two or more surface that do not contain pulp involvement

Exclusion Criteria:

* did not attend their follow-up appointments

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Crown success | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  Crown success was categorized as "successful" if no loss or fractures occurred and "unsuccessful" otherwise. Failed cases are classified as decementation, occlusal wear and fracture. Fracture classification includes large loss and chipped cases.

SECONDARY OUTCOMES:
Plaque Index | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  The Plaque Index scores of all teeth, including those treated with crowns (FGC group) and their symmetrical, healthy counterparts (control group), were evaluated and recorded, both before and after the application of the fiberglass crowns. The plaque Index was evaluated using the criteria established by Silness and Löe, with scores assigned as follows; 0 (the best): no plaque, 1: a film of plaque adhering to the free gingival margin and adjacent area of the tooth, 2: moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye and, 4 (the worst): abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin. In the evaluation of the periodontal index, plaque control was carried out by utilizing a plaque-disclosing agent.
Gingival Index | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  The Gingival Index scores of all teeth, including those treated with crowns (FGC group) and their symmetrical, healthy counterparts (control group), were evaluated and recorded, both before and after the application of the fiberglass crowns. The Gingival Index was evaluated using the criteria established by Silness and Löe, with scores assigned as follows; 0 (the best): normal gingiva, 1: mild inflammation, 2: moderate inflammation, and 4 (the worst): severe inflammation.

OTHER OUTCOMES:
Parental Satisfaction with fiberglass crown restorations | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  Parental satisfaction was assessed for appearance, color, shape, size, and durability according to Roberts et al.'s criteria. A 1-5 scale was used with 1=very dissatisfied and 5=very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfikar Zahit Ciftci, Phd, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)